CLINICAL TRIAL: NCT04656002
Title: As a Second-line Treatment for Metastatic Gastric Adenocarcinoma Patients, the Safety and Effective of Vactosertib Administration in Combination With Paclitaxel+Ramucirumab is Evaluated, and a Phase 2a Clinical Trial to Biomarkers
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Seung tae Kim,PhMD, PH,MD, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-05-175
Record Dates: First submitted 2020-11-30; First posted 2020-12-07 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — vactosertib

STUDY DESIGN:
Intervention Model Description: TEW-7197 300 mg BID 5D on/2D off
  + Ramucirumab IV 8 mg/kg every 2weeks +Paclitaxel 80 mg/m2 day1.8.15 every 28days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Paclitaxel, Ramucirumab + TEW-7197 (Experimental): Take Baektoseotip (TEW-7197) twice a day for 5 days and take a break for 2 days (5D on/2D off). With this method, progression up to the 28th day is taken as one cycle. Take it with or without food every twelve hours
  -Paclitaxel, Ramucirumab Intravenous (IV) Ramucirumab injection, provided as a single-use 500-mg/50-mL vial containing 10 mg/mL of product in histidine buffer, with disease progression, toxicity requiring discontinuation, or without interruption for any reason. After diluting to 8 mg/kg every 2 weeks, IV It is administered by infusion.
  Paclitaxel is administered at a dose of 80 mg/m2 on days 1, 8 and 15 of a 28-day cycle, with disease progression, toxicity requiring discontinuation, or without interruption for any reason.
  Interventions: Drug: Vactosertib

INTERVENTIONS:
Drug: Vactosertib — Take Baektoseotip (TEW-7197) twice a day for 5 days and take a break for 2 days (5D on/2D off). With this method, progression up to the 28th day is taken as one cycle. Take it with or without food every twelve hours
  Other Names: TEW-7197

SUMMARY:
This clinical trial is to evaluate the efficacy and safety of subjects with metastatic gastric adenocarcinoma or adenocarcinoma of the gastroesophageal junction. In addition, this clinical trial is performed to analyze the genome-specific response rate and genome analysis to identify predictive markers that respond to investigational drug administration.

DETAILED DESCRIPTION:
4 weeks (28 days) administration is considered as 1 cycle.

[Bactosertib／TEW-7197] A 300mg dose is administered orally as tablets twice a day for 5 days, followed by a 2 day holiday. (5 days medication/2 days off). All doses are taken in the morning/evening, approximately 12 hours apart, regardless of food.

[Ramucirumab (ramucirumab)] A dose of 8 mg/kg (8 mg per kg of body weight) is administered once for 60 minutes at the 1st and 15th days of each cycle. This drug is administered directly into a blood vessel using an infusion pump.

[paclitaxel (paclitaxel)] A dose of 80mg/m2 is administered intravenously for 60 minutes at the 1st, 8th, and 15th days of each cycle and is withdrawn for 1 week.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically or cytologically confirmed gastric cancer, including gastric adenocarcinoma or GEJ adenocarcinoma.
2. Patients with metastatic or locally recurrent unresectable disease.
3. Patients with diseased lesions that can be measured using standard computed tomography (CT) or magnetic resonance imaging (MRI).
4. Patients who have experienced disease progression during or after primary therapy for metastatic disease.
5. Patients over 19 years of age.
6. All clinically significant toxic effects of previous chemotherapy, surgery, radiation therapy, or hormone therapy are rated ≤1 (or neuropathic Cases ≤2 grade) (excluding hair loss).
7. Patients with an Eastern Oncology Cooperative Group Performance Status (ECOG PS) score of 0 or 1.
8. Total bilirubin ≤1.5 mg/dL (25.65 µmol/L), and aspartic acid aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3.0 x upper limit of normal (ULN; or 5.0 x with liver metastasis) Patients with adequate liver function as defined by ULN).

etc

Exclusion Criteria:

1. Patients previously receiving treatment targeting the TGF-β signaling pathway
2. Patients who previously received Taxane-based chemotherapy
3. Patients with recorded and/or symptomatic brain or meningeal metastases.
4. Patients who experienced Grade 3-4 GI bleeding within 3 months prior to enrollment.
5. Patients who have experienced arterial thromboembolic events including, but not limited to, myocardial infarction, transient ischemic attack, cerebrovascular attack, or unstable angina within 6 months prior to enrollment.
6. Ongoing or active infection, symptomatic congestive heart failure, unstable angina, symptomatic or poorly controlled cardiac arrhythmias, uncontrolled thrombotic or hemorrhagic disease, interstitial pneumonia or pulmonary fibrosis, or in the judgment of the treating physician. Patients with other serious medical conditions that are not controlled.
7. Patients with ongoing or active psychiatric conditions or social situations that may limit adherence to treatment.
8. Patients with uncontrolled or poorly controlled hypertension (systolic >160 mmHg or diastolic >100 mmHg for >4 weeks) despite standard medical care.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | up to 24momths

SECONDARY OUTCOMES:
Disease control rate | up to 24momths

CONTACTS AND LOCATIONS:
Overall Officials: SeungTae Kim, PhMD, Principal Investigator — Samsung Medical Center